CLINICAL TRIAL: NCT02595047
Title: Phase 1/2 Study of Autologous Tissues/Body Surface Organs Prefabrication in Tissue Reconstruction
Brief Title: Autologous Prefabrication of Body Surface Tissues/ Organs(e.g. Joint)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-Feng Li, MD, PhD, Professor, Head of the Department of Plastic and Reconstructive Surgery, Shanghai 9th People'sHospital Affiliation: Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2012]23
Record Dates: First submitted 2015-09-27; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Soft Tissue Infections; Intentional Self Harm by Other Specified Means
Keywords: Self-regeneration, in vivo tissue prefabrication,
MeSH Terms: conditions — Soft Tissue Infections | interventions — Histocompatibility Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tissue/ organ prefabrication (Experimental): in vivo generation of autologous tissue for joint replacement
  Interventions: Procedure: tissue/ organ prefabrication

INTERVENTIONS:
Procedure: tissue/ organ prefabrication — tissue/ organ is prefabricated in vivo independent of exogenous factors for replacement/ reconstruction purposes
  Other Names: ear, joint, bone, cartilage

SUMMARY:
The purpose of this study is to observe the feasibility and its application of autologous prefabrication for body surface tissues/oranges

DETAILED DESCRIPTION:
In the field of tissue regeneration techniques, the in vitro processes and other exogenous factors still have many uncertainties. These uncertainties have hampered road to the clinical application. As the importance of in vivo environment has aroused more awareness, the investigators validated the hypothesis that the feasibility of self-regeneration prefabricated unaided by any in vitro culture process or exogenous elements.

ELIGIBILITY:
Inclusion Criteria:

* With body surface tissue or organ defects (e.g., ear, nose, bone and joint) requiring reconstruction.

Exclusion Criteria:

* evidence of infection, ischemia, ulcer or other pathological changes within the prefabricated area which defined as not suitable for tissues regeneration
* history of delayed healing, radiational therapy;
* significant renal, cardiovascular, hepatic and psychiatric diseases;
* significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV);
* BMI >30;
* history of any hematological disease, including leukopenia, thrombocytopenia, or thrombocytosis;
* Evidence of malignant diseases
* unwillingness to participate.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of major adverse events | through study completion 12 months after prefabrication
  Including infection, necrosis, resorption

SECONDARY OUTCOMES:
Feasibility of self-prefabrication | 3, 6, and 12 months after prefabrication
  To observe the regeneration changes of prefabricated neo-tissue by histology (staining) and biomechanical analysis (bone density, Young's modulus)

OTHER OUTCOMES:
survival of prefabricated tissue after grafting | 3, 6, 12, and 36 months after grafting
  Assessed by radiologic imaging (CT, MRT)
biomechanical function of prefabricated tissue after grafting | 3, 6, 12, and 36 months after grafting
  Assessed by total range of motion (degree)
biomechanical function of prefabricated tissue after grafting | 3, 6, 12, and 36 months after grafting
  Assessed by grip strength (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Li, MD,PhD, Study Director — Department of Plastic and Reconstructive Surgery, Shanghai 9th People'sHospital
Locations (1):
- Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China